CLINICAL TRIAL: NCT05845138
Title: An Open-Label, Multi-center Phase Ⅰb/Ⅱ Study of SHR-A1811 Combined With Capecitabine in Treatment of Unresectable or Metastatic Breast Cancer With Low HER2 Expression.
Brief Title: A Study of SHR-A1811 Combined With Capecitabine in Treatment of Unresectable or Metastatic Breast Cancer With Low HER2 Expression.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-207
Record Dates: First submitted 2023-04-18; First posted 2023-05-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Capecitabine

STUDY DESIGN:
Intervention Model Description: SHR-A1811 combined with capecitabine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 combined with capecitabine (Experimental)
  Interventions: Drug: SHR-A1811 for injection ; capecitabine

INTERVENTIONS:
Drug: SHR-A1811 for injection ; capecitabine — SHR-A1811 for injection; Capecitabine tablets

SUMMARY:
The study is being conducted to evaluate the safety, tolerability， preliminary efficacy, pharmacokinetics, and immunogenicity of SHR-A1811 combined with capecitabine in treatment of unresectable or metastatic breast cancer with low HER2 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 (inclusive).
2. HER2 low expression unresectable or metastatic breast cancer confirmed by histology or cytology.
3. ECOG score is 0 or 1.
4. An expected survival of ≥ 12 weeks.
5. At least one measurable lesion according to RECIST v1.1 criteria.
6. Women of childbearing potential (WOCBP) subjects must agree to use highly effective contraception for 7 months from the start of study screening until the last study medication and agree not to breastfeeding.
7. Patients voluntarily joined the study and signed informed consent, had good compliance and willingness to cooperate with the visit and study related procedures.

Exclusion Criteria:

1. Have other malignancies within the past 5 years.
2. Presence with uncontrollable third space effusion.
3. Have surgical treatment, radiotherapy, chemotherapy, immunotherapy, molecular targeted therapy, biological therapy or other drug clinical studies within 4 weeks before the first medication.
4. Accepted antibody drug conjugates containing etoisomercan derivative topoisomerase I inhibitor.
5. Clinically significant cardiovascular disorders.
6. Presence of active hepatitis B, hepatitis C, cirrhosis,or serious infected persons requiring antibiotic, antiviral or antifungal control.
7. The toxicity from previous anti-tumor treatment has not recovered to ≤ grade I.
8. Known to be allergic to any study drug or any of its excipients, or to humanized monoclonal antibody products.
9. Failure to swallow, chronic diarrhea, intestinal obstruction, or presence of other factors affecting drug administration and absorption.
10. Presence of other serious physical or mental diseases or laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT（Phase I (dose exploration phase) ） [ Time Frame: 21 days after the first administration of each subject ] | 21 days after the first administration of each subject ]
Incidence of AEs（Phase I (dose exploration phase) ） | from Day1 to 40 days after last dose
Incidence of SAEs（Phase I (dose exploration phase) ） | from Day1 to 40 days after last dose
Objective response rate（Phase II (efficacy expansion phase)） | One year after the last subject was enrolled in the group

SECONDARY OUTCOMES:
Duration of response(DoR ) | One year after the last subject was enrolled in the group
Progression Free Survival(PFS) | One year after the last subject was enrolled in the group
Objective response rate（Phase I (dose exploration phase)） | One year after the last subject was enrolled in the group
Incidence of AEs（Phase II (efficacy expansion phase)） | from Day1 to 40 days after last dose
Incidence of SAEs（Phase II (efficacy expansion phase)） | from Day1 to 40 days after last dose

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijng
  - Guangxi Medical University Affiliated Tumor Hospital & Oncology Medical College, Nanning, Guangxi
  - Shantou Central Hospital, Shantou, Guangzhou
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital&Institute, Jinan, Shandong
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided